CLINICAL TRIAL: NCT06299397
Title: The Effect of Breastfeeding Education and Humor-Based Practices on Breastfeeding Motivation and Attachment in the Antenatal Period
Brief Title: Breastfeeding Education and Humor-Based Practices on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Inonu-SBF-4
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Humor as Topic; Breast Feeding; Mother-Child Relations; Breastfeeding, Exclusive
Keywords: humor as topic; breastfeeding; bonding; antenatal; motivation
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants determined by the researchers before starting the study were divided into experimental and control groups by randomization method. Humor-based breastfeeding education was given to women in the experimental group for 35-45 minutes once a week for 2 weeks on specified days and hours. Breastfeeding education was given in practice. Then, humor was practiced with songs and clown costumes. An interim test was administered one month after this application and a final test was administered three months later.
Who Masked: Participant, Investigator
Masking Description: After randomization was performed by a researcher independent of the study, it was decided by lottery method which group would be the experiment and which group would be the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding-Humor group (Experimental): 32 pregnant women were included in the experimental group determined by randomization method. Consent to participate in the study was obtained from these pregnant women. After obtaining consent, a pre-test was conducted. Afterwards, pregnant women were given breastfeeding education and humor practice. The application was applied once a week, twice a week. An interim test was administered 1 month after the application, and a final test was administered 3 months later.
  Interventions: Behavioral: breastfeeding - humor training
- Control Group (Sham Comparator): After randomization, consent was obtained from the pregnant women determined that they agreed to participate in the study. The pregnant women in the control group were given a pre-test before starting the study, an interim test 1 month after the start, and a final test 3 months later.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: breastfeeding - humor training — Breastfeeding and humor-based practice will continue for 35-45 minutes, once a week for 2 weeks.
  Arms: Breastfeeding-Humor group
Other: Control Group — After randomization, consent was obtained from the pregnant women determined that they agreed to participate in the study. The pregnant women in the control group were given a pre-test before starting the study, an interim test 1 month after the start, and a final test 3 months later.
  Arms: Control Group

SUMMARY:
The aim of this study is to determine the effect of breastfeeding education and humor-based practices in the antenatal period on breastfeeding motivation and attachment. 32-36 patients who applied to Bartın Gynecology and Children's Hospital for the project. It will consist of 64 pregnant women (32 experimental and 32 control group) at gestational week. Pregnant women who agree to participate in the project between these months will receive 30-45 minutes of humor practice after 30 minutes of breastfeeding training in the first session. The education and humor application will be implemented again a week later, on the same day, at the same time and in the same place. In the humor application, dance performances, applause, singing and laughter accompanied by 5 songs determined by the researchers will be included. The training program prepared for breastfeeding education will be applied to pregnant women. Then, humor will be applied. A pre-test will be administered before the training, a mid-test 1 month after the training, and a post-test in the 3rd month. Project data will be collected using the 'Introductory Information Form', 'Breastfeeding Motivation Scale' and 'Maternal Attachment Scale'.

DETAILED DESCRIPTION:
Breastfeeding is the ideal source of nutrition for babies. The World Health Organization (WHO) recommends continuing breastfeeding exclusively with breast milk for the first 6 months and with complementary foods for up to 3 years. Breastfeeding is extremely effective on the health of the baby and mother. The aim of this study is to determine the effect of breastfeeding education and humor-based practices in the antenatal period on breastfeeding motivation and attachment. 32-36 patients who applied to Bartın Gynecology and Children's Hospital for the project. It will consist of 64 pregnant women (32 experimental and 32 control group) at gestational week. Pregnant women who agree to participate in the project between these months will receive 30-45 minutes of humor practice after 30 minutes of breastfeeding training in the first session. The education and humor application will be implemented again a week later, on the same day, at the same time and in the same place. In the humor application, dance performances, applause, singing and laughter accompanied by 5 songs determined by the researchers will be included. The training program prepared for breastfeeding education will be applied to pregnant women. Then, humor will be applied. A pre-test will be administered before the training, a mid-test 1 month after the training, and a post-test in the 3rd month. Project data will be collected using the 'Introductory Information Form', 'Breastfeeding Motivation Scale' and 'Maternal Attachment Scale'.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Having a healthy pregnancy,
* Being literate,
* 32-36. Being in the gestational week,
* Being primiparous,
* Not having any psychiatric diagnosis.

Exclusion Criteria:

* Not having attended one of the trainings
* incompletely filling out the questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Being pregnant in the primiparous period
Enrollment: 64 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Motivation Scale | 3 month
  The scale consists of 24 items and 5 sub-dimensions. Subdimensions of the scale; They were determined as intrinsic motivation, integrated regulation, identified regulation, introjected regulation, and external regulation. Scale items are rated between 'I strongly disagree' (1 point) and 'I strongly agree' (4 points). The scale is a 4-point Likert type, and each item receives a score between 1 and 4. The total score of the scale is not calculated. The score of the sub-dimensions is calculated by taking the average of the scale sub-dimension scores. It has been stated that the higher the score received from the scale sub-dimension, the higher the motivation representing that sub-dimension

SECONDARY OUTCOMES:
Maternal Attachment Scale | 3 month
  It is a 26-item 4-point Likert type scale, with each item ranging from "always" to "never". Each item contains direct statements and is calculated as Always (a) = 4 points, Often (b) = 3 points, Sometimes (c) = 2 points and Never (d) = 1 point. An overall score is obtained from the sum of all items. A high score indicates high maternal attachment. The lowest score obtained from the scale varies between 26 and the highest score 104. The scale has no cut-off score.

CONTACTS AND LOCATIONS:
Overall Officials: Simge Ozturk, Ph.D, Principal Investigator — Bartın Unıversity
Locations (1):
- Simge OZTURK, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No